CLINICAL TRIAL: NCT04345016
Title: Remote Monitoring of Healed Diabetic Foot Ulcers With Podimetrics Temperature Monitoring System for Prevention of Diabetic Foot Ulcers
Brief Title: Impact of Remote Foot Temperature Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Mid-Atlantic Permanente Medical Group, P.C. (Unknown); Podimetrics, Inc. (Industry); Mid-Atlantic Permanente Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MA-16-134
Record Dates: First submitted 2020-04-07; First posted 2020-04-14 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Foot Ulcer, Diabetic
Keywords: diabetic foot; diabetic foot ulcer; prevention; resource utilization; foot temperature monitoring; telemedicine
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The investigators evaluated diabetic foot-related outcomes and associated resource utilization for each participant during three distinct phases: the two years before study participation, the one year during the foot temperature monitoring intervention, and the period after the intervention ended through the date of the analysis (January, 2020).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All Participants (Experimental): Eligible participants were provided a once-daily remote foot temperature monitoring mat (Podimetrics SmartMat; Podimetrics Inc., Somerville MA) during the intervention/treatment phase. Each was followed for one year or until study disenrollment, health plan disenrollment, death, or end of the study and follow-up period. Outcomes data from eligible participants from the two years prior to the intervention/treatment phase and the period of time after the intervention ended through the analysis date (2020-01-01) were evaluated. For this period, these participants received standard medical and diabetic foot care.
  Interventions: Device: Once-daily remote foot temperature monitoring

INTERVENTIONS:
Device: Once-daily remote foot temperature monitoring — Participants were provided a once-daily remote foot temperature monitoring mat (Podimetrics SmartMat; Podimetrics Inc., Somerville MA) which they used for one year or until dying, dropping out of the study, or disenrolling at a member of the health plan administering the study.

SUMMARY:
One of the only evidence-based practices for the prevention of diabetic foot ulcer recurrence is once-daily foot temperature monitoring, which is recommended by multiple clinical practice guidelines for high-risk patients, including those with history of foot ulcers. The purpose of this research study is to evaluate the use of once-daily foot temperature monitoring to reduce the occurrence and recurrence of diabetic foot ulcers and reduce total health care utilization for diabetic patients with a foot ulcer that has healed in the past 24 months.

DETAILED DESCRIPTION:
Skin temperature monitoring as a useful tool to detect tissue at risk for breakdown and ulceration first emerged in the 1970s and has been examined by several investigators. For neuropathic wounds (excluding acute injury) the hypothesized mechanism is believed to be repetitive stress and micro-trauma leading to enzymatic autolysis of tissue, inflammation, and a resulting measurable increase in local skin temperature.

In 1997, a paper was published examining 143 consecutive patients presenting to the University of Texas' High Risk Diabetic Foot Clinic. They hypothesized that individuals with acute pathology would show an increase in skin temperature when comparing the affected foot to the contralateral unaffected foot. Mean delta-temperatures for neuropathic ulcers and Charcot arthropathy were found to be 5.6°F (n=44, p<0.0001) and 8.3°F (n=21, p<0.0001), respectively. No statistical difference was found in neuropathic participants without acute pathology (n=78).

In a project funded by the National Institute of Health, the same investigators conducted a series of studies, published between 2004 and 2007, examining the impact of self-assessed dermal thermometry in high-risk diabetic patients In the first randomized controlled trial in 2004, 85 patients were assigned to one of two groups, Usual Therapy or Enhanced Therapy.

Participants were eligible if they had either a history of foot ulceration or lower extremity amputation, or if they had moderate to severe peripheral sensory neuropathy with a foot deformity. Both groups received therapeutic footwear, diabetic education, and regular foot evaluation by a podiatrist. Enhanced Therapy participants additionally received a hand-held dermal thermometer to self-record dermal temperatures at six sites on each foot, twice per day. If a delta-temperature between any two corresponding sites was found to be greater than 4 F, participants were instructed to reduce activity and contact the study nurse. After six months of follow-up, Enhanced Therapy participants experienced significantly fewer foot ulcerations and Charcot fractures (2% vs. 20%, p=0.01) than the Usual Therapy group. The study was blinded to physician only. A limitation of the study was the difficulty in determining whether the Enhanced Therapy group received greater attention by the care team, and therefore better monitoring and therapy.

In their second randomized controlled trial conducted in 2007, 173 participants were enrolled between the Texas A&M University Health Science Center and the Rosalind Franklin University of Medicine and Science. Participants were eligible if they were diabetic and had a history of previous foot ulcer, and were assigned to one of three groups: Standardized Therapy, Structured Foot Exam, and Enhanced Therapy. All three groups received standard of care (therapeutic footwear, diabetic foot education, and regular foot evaluation by a podiatrist) and were instructed to contact the study nurse if they noticed any abnormalities during their daily foot inspection. The Structured Foot Exam group, in addition to standard training, were instructed to conduct a structured foot inspection twice daily with the assistance of a mirror and record any noted changes in color, swelling or warmth in a detailed log book. The Enhanced Therapy group, in addition to standard training, were trained to use a hand-held dermal thermometer to record daily foot temperatures at the six locations on each foot, noting any delta-temperatures between feet. Should a difference between corresponding sites be found greater than 4 degF for two consecutive days, participants were instructed to contact the study nurse and decrease activity until temperatures normalized. After 15 months of follow-up, Enhanced Therapy participants had fewer foot ulcers than Standard Therapy participants and Structured Foot Examination participants (Enhanced Therapy 8.5% vs. Standard Therapy 29.3%, p=0.0046; and Enhanced Therapy 8.5% vs. Structured Foot Examination 30.4%, p=0.0029). No difference was found between Standard Therapy and Structured Foot Exam groups. The study was physician blinded as before.

In the third RCT, 225 patients from the Southern Arizona VA Healthcare System (Tucson, AZ) were randomized between the Standard Therapy Group and the Dermal Thermometry Group. Eligible participants had either a history of foot ulcer or partial foot amputation or a history of neuropathy and structural foot deformity or limited joint mobility. Participants were followed for 18 months, blinded to the physician. Both groups received standard of care and performed daily structured foot self-examinations. The Dermal Thermometry Group additionally received a hand-held dermal thermometer to assess six plantar foot sites twice per day. Dermal Thermometry Group patients were instructed to contact the study nurse if delta-temperature between corresponding locations on the feet exceeded 4 F for two consecutive days and decrease activity until the temperature asymmetry normalized. Dermal Thermometry patients were 61% less likely to ulcerate: 12.2% ulceration in the Standard Therapy Group vs. 4.7% ulceration in the Dermal Thermometry Group (O.R. 3.0, 95% CI 1.0-8.5, p=0.038). Further, proportional hazards regression analysis adjusting for elevated foot ulcer classification (International Working Group Risk Factor 3), age, and minority status suggested that temperature-guided avoidance therapy was associated with a significantly longer time to ulceration (p = 0.04).

One significant challenge to temperature guided avoidance therapy owe to the manual process of collecting and recording temperatures. With current technologies the following steps must be taken each day: temperatures measurements are acquired at six different locations on each foot, the values are recorded in an organized fashion in a log book, and the history of values are interpreted for trends in temperature difference between each foot. This process places a significant burden on the patient. Further, as day-to-day usage of the technology cannot be tracked, managing adherence becomes challenging.

The purpose of this study is to demonstrate the feasibility of temperature-guided avoidance therapy via the a foot temperature monitoring telemedicine mat (Podimetrics SmartMat; Podimetrics Inc., Somerville MA) on preventing the occurrence of diabetic foot ulcers and associated resource utilization in patients with a recently healed diabetic foot ulcer.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of diabetes mellitus (type 1 or 2)
* a history of diabetic foot ulcer or amputation which healed within the 24 months prior to enrollment
* adequate lower extremity vascular supply, defined as presence of palpable bilateral posterior tibial and dorsalis pedis pulses or an ankle brachial index exceeding 0.5 documented within the 12 months preceding study enrollment
* the ability to provide informed consent

Exclusion Criteria:

* baseline inflammatory foot conditions, including unhealed ulcer or lesion (dorsal or plantar), active Charcot arthropathy, ongoing foot infection, or ongoing cellulitis
* a history of amputation more proximal than a transmetatarsal amputation in either foot
* inability to ambulate without the assistance of a wheelchair, walker, or crutches
* travel plans expected to interrupt the use of the study device for longer than two consecutive weeks
* any condition which, in the investigator's judgment, rendered the patient unsuitable or unreliable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
rate of diabetic foot ulcer recurrence in before phase of trial | From two years before the date of enrollment until the date of enrollment, exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of new diabetic foot ulcers occurring to participants (total number of diabetic foot ulcers divided by the total exposure duration for the participants)
rate of diabetic foot ulcer recurrence in during phase of trial | From the date of enrollment until the participant completed one year using the study device, or until withdrawing consent, dropping out, dying, or disenrolling as a beneficiary of the health plan sponsoring the trial
  temporal rate of new diabetic foot ulcers occurring to participants (total number of diabetic foot ulcers divided by the total exposure duration for the participants)
rate of diabetic foot ulcer recurrence in after phase of trial | From completing use of the study device until the analysis date on Jan 1, 2020 (between six months and three years on average for participants), exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of new diabetic foot ulcers occurring to participants (total number of diabetic foot ulcers divided by the total exposure duration for the participants)

SECONDARY OUTCOMES:
adherence in daily use of the study device | From the date of enrollment until the participant completed one year using the study device, or until withdrawing consent, dropping out, dying, or disenrolling as a beneficiary of the health plan sponsoring the trial
  total number of uses during each unique day during the intervention divided by the total number of exposure days during the treatment phase of the study
rate of inflammation episodes detected by the study device | From the date of enrollment until the participant completed one year using the study device, or until withdrawing consent, dropping out, dying, or disenrolling as a beneficiary of the health plan sponsoring the trial
  total number of times the study device identified inflammation to participants during the treatment phase of the study divided by the total number of exposure days during the treatment phase of the study
rate of severe diabetic foot ulcer recurrence in before phase of trial | From two years before the date of enrollment until the date of enrollment, exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of new diabetic foot ulcers with classification > UT-1A on the University of Texas grading system occurring to participants (total number of diabetic foot ulcers with classification > UT-1A divided by the total exposure duration for the participants)
rate of severe diabetic foot ulcer recurrence in during phase of trial | From the date of enrollment until the participant completed one year using the study device, or until withdrawing consent, dropping out, dying, or disenrolling as a beneficiary of the health plan sponsoring the trial
  temporal rate of new diabetic foot ulcers with classification > UT-1A on the University of Texas grading system occurring to participants (total number of diabetic foot ulcers with classification > UT-1A divided by the total exposure duration for the participants)
rate of severe diabetic foot ulcer recurrence in after phase of trial | From completing use of the study device until the analysis date on Jan 1, 2020 (between six months and three years on average for participants), exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of new diabetic foot ulcers with classification > UT-1A on the University of Texas grading system occurring to participants (total number of diabetic foot ulcers with classification > UT-1A divided by the total exposure duration for the participants)
rate of inpatient admissions in before phase of trial | From two years before the date of enrollment until the date of enrollment, exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of hospital admissions (total number of hospitalizations divided by the total exposure duration for the participants)
rate of inpatient admissions in during phase of trial | From the date of enrollment until the participant completed one year using the study device, or until withdrawing consent, dropping out, dying, or disenrolling as a beneficiary of the health plan sponsoring the trial
  temporal rate of hospital admissions (total number of hospitalizations divided by the total exposure duration for the participants)
rate of inpatient admissions in after phase of trial | From completing use of the study device until the analysis date on Jan 1, 2020 (between six months and three years on average for participants), exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of hospital admissions (total number of hospitalizations divided by the total exposure duration for the participants)
rate of outpatient visits in before phase of trial | From two years before the date of enrollment until the date of enrollment, exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of outpatient visits (any department/specialty) (total number of outpatient visits divided by the total exposure duration for the participants)
rate of outpatient visits in during phase of trial | From the date of enrollment until the participant completed one year using the study device, or until withdrawing consent, dropping out, dying, or disenrolling as a beneficiary of the health plan sponsoring the trial
  temporal rate of outpatient visits (any department/specialty) (total number of outpatient visits divided by the total exposure duration for the participants)
rate of outpatient visits in after phase of trial | From completing use of the study device until the analysis date on Jan 1, 2020 (between six months and three years on average for participants), exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of outpatient visits (any department/specialty) (total number of outpatient visits divided by the total exposure duration for the participants)
rate of lower extremity amputations in before phase of trial | From two years before the date of enrollment until the date of enrollment, exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of lower extremity amputations (total number of amputations divided by the total exposure duration for the participants)
rate of lower extremity amputations in during phase of trial | From the date of enrollment until the participant completed one year using the study device, or until withdrawing consent, dropping out, dying, or disenrolling as a beneficiary of the health plan sponsoring the trial
  temporal rate of lower extremity amputations (total number of amputations divided by the total exposure duration for the participants)
rate of lower extremity amputations in after phase of trial | From completing use of the study device until the analysis date on Jan 1, 2020 (between six months and three years on average for participants), exclusive of periods when the participant was not a beneficiary of the health plan sponsoring the trial
  temporal rate of lower extremity amputations (total number of amputations divided by the total exposure duration for the participants)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Isaac, DPM, Principal Investigator — Kaiser Permanente Mid-Atlantic States Mid-Atlantic Permanente Medical Group
Locations (3):
- United States (3):
  - Kensington Medical Center, Kensington, Maryland
  - Largo Medical Center, Upper Marlboro, Maryland
  - Springfield Medical Center, Springfield, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request for research purposes by request to the Study Official (Adam Isaac, DPM) contingent upon approval by Kaiser Permanente Mid-Atlantic Permanente Research Institute.
Supporting Information: Analytic Code
Time Frame: Data will be available beginning after peer review and publication.
Access Criteria: Data may be used for research purposes only. No commercial use permitted. It is available upon reasonable request of the Study Official (Adam Isaac, DPM) contingent upon approval by Kaiser Permanente Mid-Atlantic Permanente Research Institute.

REFERENCES:
- [Background] Lavery LA, Higgins KR, Lanctot DR, Constantinides GP, Zamorano RG, Athanasiou KA, Armstrong DG, Agrawal CM. Preventing diabetic foot ulcer recurrence in high-risk patients: use of temperature monitoring as a self-assessment tool. Diabetes Care. 2007 Jan;30(1):14-20. doi: 10.2337/dc06-1600. PMID 17192326
- [Background] Lavery LA, Higgins KR, Lanctot DR, Constantinides GP, Zamorano RG, Armstrong DG, Athanasiou KA, Agrawal CM. Home monitoring of foot skin temperatures to prevent ulceration. Diabetes Care. 2004 Nov;27(11):2642-7. doi: 10.2337/diacare.27.11.2642. PMID 15504999
- [Background] Gordon IL, Rothenberg GM, Lepow BD, Petersen BJ, Linders DR, Bloom JD, Armstrong DG. Accuracy of a foot temperature monitoring mat for predicting diabetic foot ulcers in patients with recent wounds or partial foot amputation. Diabetes Res Clin Pract. 2020 Mar;161:108074. doi: 10.1016/j.diabres.2020.108074. Epub 2020 Feb 25. PMID 32109516
- [Background] Frykberg RG, Gordon IL, Reyzelman AM, Cazzell SM, Fitzgerald RH, Rothenberg GM, Bloom JD, Petersen BJ, Linders DR, Nouvong A, Najafi B. Feasibility and Efficacy of a Smart Mat Technology to Predict Development of Diabetic Plantar Ulcers. Diabetes Care. 2017 Jul;40(7):973-980. doi: 10.2337/dc16-2294. Epub 2017 May 2. PMID 28465454
- [Background] Banks JL, Petersen BJ, Rothenberg GM, Jong AS, Page JC. Use of a Remote Temperature Monitoring Mat for the Early Identification of Foot Ulcers. Wounds. 2020 Feb;32(2):44-49. PMID 32155121
- [Background] Killeen AL, Brock KM, Dancho JF, Walters JL. Remote Temperature Monitoring in Patients With Visual Impairment Due to Diabetes Mellitus: A Proposed Improvement to Current Standard of Care for Prevention of Diabetic Foot Ulcers. J Diabetes Sci Technol. 2020 Jan;14(1):37-45. doi: 10.1177/1932296819848769. Epub 2019 May 23. PMID 31122064
- [Background] Killeen AL, Walters JL. Remote Temperature Monitoring in Diabetic Foot Ulcer Detection. Wounds. 2018 Apr;30(4):E44-E48. PMID 29718822
- [Derived] Isaac AL, Swartz TD, Miller ML, Short DJ, Wilson EA, Chaffo JL, Watson ES, Hu H, Petersen BJ, Bloom JD, Neff NJ, Linders DR, Salgado SJ, Locke JL, Horberg MA. Lower resource utilization for patients with healed diabetic foot ulcers during participation in a prevention program with foot temperature monitoring. BMJ Open Diabetes Res Care. 2020 Oct;8(1):e001440. doi: 10.1136/bmjdrc-2020-001440. PMID 33055233